CLINICAL TRIAL: NCT06870539
Title: Feasibility of Saliva and Remote Monitoring of Active Cytomegalovirus (CMV) Infection and Symptoms During Ovarian Cancer Treatment
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 24-011332; NCI-2025-01230 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-011332 (Other: Mayo Clinic Institutional Review Board); P50CA136393 (NIH)
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Cancer-related Cognitive Dysfunction; Cytomegaloviral Infection; Fallopian Tube Carcinoma; Ovarian Carcinoma; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Cytomegalovirus Infections; Fallopian Tube Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples retained for future research only with permission of participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo saliva sample collection as well as in-clinic or at-home blood sample collection on study. Patients also complete questionnaires, undergo cognitive function testing, and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
This study evaluates the feasibility and accuracy of using saliva to remotely monitor cytomegalovirus (CMV) infection in individuals receiving treatment for ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Ability to read and write in English
* Diagnosed with ovarian cancer (ovarian, primary peritoneal, fallopian tube)
* Receiving care from providers at Mayo Clinic
* Regardless of diseases status, actively receiving treatment for ovarian cancer (frontline, maintenance, progression, recurrence)

Exclusion Criteria:

* Pregnant at the time of study participation
* Inability to provide informed written consent
* History of dementia, stroke, brain tumors or other condition which may impair cognitive functioning

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ovarian cancer undergoing active treatment at the Mayo Clinic
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Using saliva and blood samples to remotely monitor cytomegalovirus (CMV) infection | Baseline
  Assessed through collection and comparison of blood and saliva samples collected from individuals receiving treatment for ovarian cancer. Samples may be collected in clinic or at home following study enrollment. Saliva will be self-collected using Oragene OGR-600 kits. Blood samples will be collected at the time of another scheduled clinic blood draw (Aim 1) or at home through a home phlebotomy service (Aim 2).

CONTACTS AND LOCATIONS:
Overall Officials: Amanika Kumar, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials
- See also: University of Minnesota Medical School Clinical Trials & Studies — https://med.umn.edu/dom/research/clinical-research-and-trials